CLINICAL TRIAL: NCT02242773
Title: MRI-Guided Active Selection for Treatment of Prostate Cancer: The Miami MAST Trial
Brief Title: MRI Based Active Selection for Treatment Trial
Acronym: MAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sanoj Punnen, MD, MAS, Associate Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20140372; 1R01CA189295-01 (NIH)
Record Dates: First submitted 2014-09-13; First posted 2014-09-17 (Estimated); Results first posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
Keywords: Active Surveillance; MRI-Guided Biopsy; Multi-parametric MRI; MP-MRI
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Active Surveillance (Experimental): Participants in this group will receive a Multi-Parametric Magnetic Resonance Imaging (MP-MRI) of the prostate/pelvis and MRI-guided prostate biopsy at baseline (0-3 months from enrollment) and at the 12th, 24th and 36th month follow up.
  Interventions: Device: Multi-Parametric MRI; Device: MRI-Guided Biopsy

INTERVENTIONS:
Device: Multi-Parametric MRI — Multi-Parametric MRI
Device: MRI-Guided Biopsy — MRI-Guided Biopsy

SUMMARY:
The main purpose of this study is to determine if Magnetic Resonance Imaging (MRI), along with MRI targeted biopsy of suspicious lesions, is of value in detecting patients who would be likely to require treatment earlier.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy confirmed adenocarcinoma of the prostate within 18 months prior to enrollment;
2. Pre-enrollment prostate biopsy must consist of at least 8 cores;
3. Biopsy reviewed by a University of Miami Pathologist;
4. Serum Prostate-Specific Antigen (PSA) ≤ 20 ng/ml within 3 months of study enrollment;
5. Age ≥ 35 and ≤ 85 years;
6. Ability to understand and willingness to sign a written informed consent document;
7. Patients must agree to undergo serial multiparametric MRI and MRI-guided biopsy;
8. Patients must agree to fill out the longitudinal psychosocial questionnaires assessing health related quality of life.

Exclusion Criteria:

1. Greater than 4 cores positive, of any Gleason score, on the University of Miami (UM) review,
2. Greater than 2 cores positive for Gleason 3+4 cancer,
3. Gleason 4+3 or higher cancer in any single biopsy core.
4. Extracapsular extension suspected on digital rectal exam with confirmation on MRI. Suspicion of extracapsular extension on MRI alone is not an exclusion for study enrollment.
5. Subject is not a candidate for multiparametric MRI with contrast. Some reasons may include (but are not limited to): renal insufficiency, foreign body or pacemakers.
6. No prior pelvic radiotherapy.
7. No prior surgery to the prostate, other than transurethral procedures for benign prostatic hyperplasia (e.g., transurethral resection, green light laser treatment).
8. No concurrent, active malignancy, other than non-metastatic skin cancer of any type, superficial bladder cancer, or early stage chronic lymphocytic leukemia (well-differentiated small cell lymphocytic lymphoma) or <stage IV follicular lymphoma. If a prior malignancy is in remission for ≥ 3 years then the patient is eligible.
9. Bilateral hip replacement.

Ages: 35 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2014-11-12 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanoj Punnen, MD, MAS, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kimbel IM, Wallaengen V, Zacharaki EI, Breto AL, Algohary A, Carbohn S, Gaston SM, Soodana-Prakash N, Freitas PFS, Kryvenko ON, Castillo P, Abramowitz MC, Ritch CR, Nahar B, Gonzalgo ML, Parekh DJ, Pollack A, Punnen S, Stoyanova R. HRS Improves Active Surveillance for Prostate Cancer by Timely Identification of Progression. Acad Radiol. 2025 Apr;32(4):2081-2089. doi: 10.1016/j.acra.2024.11.008. Epub 2024 Dec 17. PMID 39694787

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Surveillance
Started | 208
Completed | 208
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Active Surveillance
Number analyzed (Participants) | 208
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 127
  >=65 years | 81
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 208
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 84
  Not Hispanic or Latino | 119
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 21
  White | 182
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 208

OUTCOME MEASURES:

1. Primary Outcome: Rate of Disease Progression Within the First Two Surveillance Biopsies
Description: The rate of disease progression among participants within the first two surveillance biopsies will be reported. Progression refers to a repeat surveillance biopsy indicating any one of the following:
  1. More than 4 positive cores involving any grade of cancer,
  2. At least two core with Gleason 3+4 cancer,
  3. Any single core with Gleason 4+3 cancer or higher,
  4. A Gleason 3+3 at diagnosis that is upgraded to Gleason 3+4, or
  5. Undergoing treatment, regardless of histological progression.
Time Frame: 24 months
Measure: Number; unit: percentage of participants
Arm/Group | Active Surveillance
Number analyzed (Participants) | 208
percentage of participants | 36.1

2. Secondary Outcome: Time-to-Biochemical Recurrence (BCR)
Description: Biochemical recurrence (BCR) is defined as prostate-specific antigen (PSA) of 0.2 or higher on two or more separate measures after surgery or an increase of nadir + 2ng/ml or more after radiation. Time-to-BCR is defined as duration in days between date of treatment and date of BCR, if BCR occurs. The investigators will follow participants who have progressed and gone on to treatment.
Time Frame: Up to 36 months
Population: Participants who underwent primary therapy for prostate cancer.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Active Surveillance
Number analyzed (Participants) | 82
days | 169 [143 to 175]

3. Secondary Outcome: Health-Related Quality of Life Scores: EPIC SF-12
Description: Health-Related Quality of Life will be assessed using scores from validated questionnaires. The Expanded Prostate Cancer Index Composite and Medical Outcomes Study Short Form-12 (EPIC SF-12) will be used to evaluate patient function and satisfaction after prostate cancer treatment. Response options for each item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing better HRQOL.
Time Frame: Up to 36 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Surveillance
Number analyzed (Participants) | 208
score on a scale
  Median score at Baseline | 31 [29 to 32]
  Median score at Last Follow-up | 31 [29 to 33]

4. Secondary Outcome: Health-Related Quality of Life Scores: MAX-PC
Description: Health-Related Quality of Life will be assessed using scores from validated questionnaires. The Memorial Anxiety Scale for Prostate Cancer (MAX-PC) will be used to measure anxiety from pre-treatment to post-treatment. The scale consists of 18 items (e.g. "I thought about prostate cancer even though I didn't mean to.") scored on a scale from 0 ("not at all") to 3 ("often"). Total scores range from 0 to 54, with higher scores indicating higher levels of anxiety.
Time Frame: Up to 36 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Surveillance
Number analyzed (Participants) | 208
score on a scale
  Median Score at Baseline | 15 [11 to 22]
  Median Score at Last Follow-up | 12 [9 to 19]

5. Secondary Outcome: Discriminative Performance of NCCN Risk and Clinical Markers for Predicting Progression on Active Surveillance
Description: The investigators will assess the incremental benefit of multiparametric MRI (mpMRI), genomic risk test, and molecular markers compared to baseline National Comprehensive Cancer Network (NCCN) risk classification for predicting progression on active surveillance. Area under the receiver operating characteristic Curve (ROC) curves produced from logistic regression modeling will be used to evaluate the performance of NCCN risk and other variables (MRI, genomic testing, and molecular markers) for predicting progression on surveillance. Participants will be categorized at baseline by NCCN risk class ranging from very low risk to intermediate risk; and into those who progressed while on the trial. Additionally, MRI results, PSA density, 4K score, and Decipher Score in combination with NCCN risk were analyzed to see their additive value on determining who will experience progression on active surveillance.
Time Frame: Up to 36 months
Measure: Number; unit: probability
Arm/Group | Active Surveillance
Number analyzed (Participants) | 208
probability
  NCCN Risk | 0.6717
  NCCN + MRI | 0.7398
  NCCN + PSA Density (PSAd) | 0.7168
  NCCN + Decipher Score | 0.6858
  NCCN + 4k Score | 0.7412

ADVERSE EVENTS:
Time Frame: Six years
Arm/Group | Active Surveillance
All-Cause Mortality (participants affected / at risk) | 2/208
Serious Adverse Events (participants affected / at risk) | 5/208
Other Adverse Events (participants affected / at risk) | 8/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Surveillance (N=208)
Hypertension (Vascular disorders) | 1 (1)
Sepsis (Infections and infestations) | 4 (4)
Urinary Tract Infection (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Surveillance (N=208)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Hematuria (Renal and urinary disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Testicular disorder (Reproductive system and breast disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-03): https://cdn.clinicaltrials.gov/large-docs/73/NCT02242773/Prot_SAP_000.pdf